CLINICAL TRIAL: NCT01985698
Title: A Single-centre, Prospective, Randomised, Controlled, Unblinded, Parallel-group Trial of Robotic-assisted Versus Laparoscopic Abdominoperineal Resection for the Curative Treatment of Low Rectal Cancer
Brief Title: A Trial of Robotic-assisted Versus Laparoscopic Abdominoperineal Resection for Treating Low Rectal Cancer
Acronym: RLAPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLAPR
Record Dates: First submitted 2013-11-09; First posted 2013-11-15 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Rectal Cancer
Keywords: Low rectal cancer; Robotic; Laparoscopic; Abdominoperineal resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robotic-assisted resection (Experimental): patients with low rectal cancer receiving robotic-assisted abdominoperineal resection.
  Interventions: Procedure: Robotic-assisted resection.
- Laparoscopic resection (Active Comparator): patients with low rectal cancer receiving laparoscopic abdominoperineal resection.
  Interventions: Procedure: Laparoscopic resection

INTERVENTIONS:
Procedure: Robotic-assisted resection. — Robotic-assisted abdominoperineal resection.
  Arms: Robotic-assisted resection
Procedure: Laparoscopic resection — Laparoscopic abdominoperineal resection
  Arms: Laparoscopic resection

SUMMARY:
In this study, the investigators assessed the difference in efficacy and safety among robotic-assisted versus laparoscopic abdominoperineal resection for patients with low rectal cancer.

DETAILED DESCRIPTION:
Patients will be eligible for inclusion if their primary tumors is low rectal cancer.

Eligible patients will be randomly assigned to robotic-assisted (arm A) versus laparoscopic (arm B) abdominoperineal resection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven rectal adenocarcinoma
* Inferior edge of the tumor located within 5 cm from the anal verge as determined by colonoscopy withdrawing and digital rectal examination
* No evidence of distant metastases (including pelvis, peritoneum, liver, lung, brain, bone, distant lymph node, etc) according to ultrasound, CT, PET-CT, etc
* Tumor assessed as cT1-T3 or ycT1-T3 after preoperative neoadjuvant chemoradiotherapy by pelvic MRI
* No other malignancies in medical history except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri
* Suitable for both robot-assisted and laparoscopic surgery
* American Society of Anesthesiologists (ASA) class I - III
* No other preoperative treatment except neoadjuvant chemoradiotherapy
* Informed consent

Exclusion Criteria:

* Tumors assessed as cT1N0 and suitable for local excision
* Signs of acute intestinal obstruction, bleeding or perforation needing emergency surgery
* More than one colorectal tumor
* Familial Adenomatosis Polyposis, Lynch Syndrome, acute inflammatory bowel disease
* Schedules need for other synchronous colon surgery
* Absolute contraindications to general anesthesia or prolonged pneumoperitoneum (ASA class > III)
* Pregnancy or lactation
* Patients and/or family members can not understand and accept this study
* Patients received chemoradiotherapy or other anti-tumor therapy before surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 30 days post operatively
  postoperative complications related to operation

SECONDARY OUTCOMES:
operative mortality | 30 days post operatively
  death occurred 30 days after operation
disease-free survival | 3 years
  disease-free survival rate at 3 years after operation
overall survival | 3 and 5 years
  overall survival rate at 3 and 5 years after operation
locoregional recurrence rate | 3 and 5 years
  local recurrence rate at 3 and 5 years after operation

OTHER OUTCOMES:
operative time | Day 1
  Time from cutting the skin to suturing the incision during the surgery, recorded in minute
rate of conversion to open surgery | Day 1
  The rate of patients actually receiving open surgery in robotic or laparoscopic surgery groups.
estimated blood loss | Day 1
  Blood loss will be measured according to the suction and the weight of wet gauze, and then minus the irrigation.
circumferential resection margin | 10 days post operatively
  The circumferential margin will be reported as "positive" or "negative" to define whether tumor is radically resected. It will be reported according to the post-operative pathology. Details are based on NCCN and Chinese guidelines for colorectal cancer.
proximal/distal resection margin | 10 days post operatively
  The proximal/distal resection margin will be reported as "positive" or "negative" to define whether tumor is radically resected. It will be reported according to the post-operative pathology. Details are based on NCCN and Chinese guidelines for colorectal cancer.
number of retrieved lymph nodes | 10 days post operatively
  It will be reported according to the post-operative pathology.
postoperative hospital stay | 30 days post operatively
  The postoperative hospital stay is defined as the number of date from the first day after operation to discharge.
self reported bladder function | at postoperative 3, 6 and 1 2 months
  This section is assessed using a self-rating scale "International prostate symptom score" (IPSS)
self reported sexual function for male patients | at postoperative 3, 6 and 1 2 months
  This section is assessed using a self-rating scale "International Index of Erectile Function" (IIEF-5).
self reported sexual function for female patients | at postoperative 3, 6 and 1 2 months
  This section is assessed using a self-rating scale "Female Sexual Function Index" (FSFI).

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Feng Q, Tang W, Zhang Z, Wei Y, Ren L, Chang W, Zhu D, Liang F, He G, Xu J. Robotic versus laparoscopic abdominoperineal resections for low rectal cancer: A single-center randomized controlled trial. J Surg Oncol. 2022 Dec;126(8):1481-1493. doi: 10.1002/jso.27076. Epub 2022 Aug 29. PMID 36036889